CLINICAL TRIAL: NCT06932718
Title: Evaluation of a Smoking Cessation Program in Workplaces in Hong Kong: a Pragmatic Randomized Controlled Trial on Mobile Phone-Based Intervention Combined With Small Incentive for Smoking Cessation
Brief Title: Smoking Cessation Programme in Workplaces in Hong Kong (Phase ⅤII)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Lok Sin Tong Benevolent Society, Kowloon (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LST SCPW P7
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Personalized chat-based support and nicotine replacement therapy sampling (NRT-S) for continued smokers at 6 months for intervention group
  Interventions: Behavioral: General health talk; Behavioral: Personalized chat-based interactions; Behavioral: Phone follow-up/counselling service; Drug: Mailed nicotine replacement therapy (NRT); Other: Small incentive
- Control (Placebo Comparator): Regular text-based support and nicotine replacement therapy sampling (NRT-S) for continued smokers at 6 months for control group
  Interventions: Behavioral: General health talk; Behavioral: Phone follow-up/counselling service; Drug: Mailed nicotine replacement therapy (NRT); Behavioral: Text message

INTERVENTIONS:
Behavioral: General health talk — Health talk provided information about hazards of tobacco (active smoking, second- and third-hand smoke), benefits of quitting smoking and methods to quit smoking.
Behavioral: Personalized chat-based interactions — Individual chat-based interactions for 3 months consist of 2 parts. The first part includes regular messages via instant messages (IM). These messages will serve as probes for real-time chat-based support in which more details explanations and motivation to encourage quitting due to financial reasons. The second part includes real-time psycho-behavioral intervention delivered by trained cessation counsellors using health economic principles on behavioral change to motivate smokers to quit. The conversation is based on participants' socio-demographic characteristics, smoking habit at baseline, and updated smoking status and mental health status assessed during online conversation and the baseline questionnaire.
  Arms: Intervention
Behavioral: Phone follow-up/counselling service — The intervention outcomes and participants' smoking status will be followed up regularly via telephone interviews (15 - 30 minutes).
Drug: Mailed nicotine replacement therapy (NRT) — Full course of NRT treatment (10 weeks) will be provided to all participants who are still smoking at 6-month follow-up and request, or willing to use NRT after advice from counsellors. Medications will be mailed from the smoking cessation clinics.
Behavioral: Text message — Regular messages will be sent twice per month within 3 months. These messages covers simple cessation advice and reminders for follow-ups.
  Arms: Control
Other: Small incentive — Positive incentive was reported to be effective in reducing smoking. Participants in the intervention group will receive HK$ 100 at 3-month follow-up. HK$ 500 will be provided to successful quitters confirmed by biochemical validation at 6 months. A total of HK$ 600 maximum will be rewarded to the participants. The amount of the incentive is comparable to other community events on smoking cessation in Hong Kong. Of note, all smokers who reported quitting, completed and passed the biochemical validation of quitting had been offered HK$ 500 in the past rounds and will also be adopted in this round.
  Arms: Intervention

SUMMARY:
Smoking cessation (SC) interventions using behavioral economics mainly focus on financial incentives, which were used to change health behaviors by utilizing a reward system to enhance long-term maintenance. Incentives have been demonstrated to enhance SC across various populations with moderate effects. Interventions for smoking cessation characterized by financial incentives focus primarily on the potential for monetary gain rather than loss. Changing the motivational strategy to combine disclosing losses with providing financial incentives may increase the effectiveness of financial consequence-based smoking cessation interventions. Thus, this study aims to test, by a 2-arm RCT, the effectiveness of an intervention of which includes mobile phone-based intervention combined with small incentive and smoking cessation in workplaces in Hong Kong; identify facilitators and barriers of successful policy implementation and quitting; examine and evaluate the company environment and their policies in promoting smoking cessation.

DETAILED DESCRIPTION:
This study will separate into two phases. Phase I is a large scale cross-sectional survey of corporations in Hong Kong to examine the employers' knowledge, attitudes and practices in promoting SC in the workplace. Phase II is a 2-arm randomized controlled trial that will be conducted to examine the effectiveness of mobile phone-based intervention combined with company health talk, brief phone counselling and nicotine replacement therapy sampling, for SC in workplaces.

Data analyses Phase I: Descriptive statistics will be used to analyze the (1) profile of the corporations, including the total number of employees and smoking employees; (2) employers/managerial staff's knowledge on smoking; (3) employers/managerial staff's attitudes on smoking cessation; (4) practices of the companies with respect to smoking cessation.

Phase II: Primary outcome is self-reported abstinence in the past 7 days at 6-month follow-up. Secondary outcomes for smoking cessation include self-reported abstinence in the past 7 days at 9- and 12-month follow-ups, the biochemically validated abstinence (defined as exhaled CO level <4ppm and saliva cotinine level ≤30 ng/ml); smoking reduction (50% or above reduction in cigarette consumption compared with baseline. Secondary outcomes for mental health include stress (Perceived Stress Scale-10), depression (Personal Health Questionnaire for Depression), anxiety (Generalized Anxiety Disorder scale) and self-rated health.

Descriptive statistics such as frequency, percentage, and mean will be used to summarize the outcomes and other variables. Chi-square tests and t-tests will be used to compare outcome variables between subgroups. The intention-to-treat (ITT) analysis will be used such that those lost to contact and refused cases at the follow-ups will be treated as no reduction in cigarette consumption nor quitting. Multiple imputations will be used to compute missing data for outcome variables. The association between intervention adherence (e.g., engagement in the IM interaction) and the primary outcome within the participants in the intervention group will be examined. The intervention effect by subgroups will be assessed respectively, including sex, age, education level, company types, previous quit attempts, cigarette dependence, and intention to quit, although the statistical power would be lower due to smaller numbers.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged 18 or above
2. Current smoking cigarettes or alternative tobacco products daily with an exhaled carbon monoxide level ≥4 ppm or a positive salivary cotinine test
3. Able to communicate in Cantonese/Mandarin and read Chinese
4. Able to use instant messaging tool (e.g. WhatsApp) for communication.
5. Stay in Hong Kong during the intervention and follow-up periods (12 months)

Exclusion Criteria:

1. Smokers who are psychologically or physically unable to communicate
2. Currently following other SC program(s)
3. Having used NRT for the past month
4. Having severe angina, serious cardiac arrhythmias and hypertension
5. Have acute myocardial event in the past month
6. Being pregnant or providing breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical validation of smoking status | 6-month
  Biochemical validated abstinence (exhaled CO level <4 ppm or a positive salivary cotinine test)

SECONDARY OUTCOMES:
Self-reported 7-day point prevalence quit rate | 1-, 3- and 12-month
  Smokers who did not smoke even a puff in the 7 days preceding the follow-up
Biochemical validation of smoking status | 12-month
  Biochemically validated quit rate (saliva cotinine level and exhale carbon monoxide test)
Self-reported reduction cigarette rate | 1-, 3-, 6- and 12-month
  Smoking reduction (50% or above reduction in cigarette consumption compared with baseline).
Self-reported use of nicotine replacement therapy (NRT) | 1-, 3-, 6- and 12-month
  Self-reported use of NRT products (e.g., gum and patches)

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No